CLINICAL TRIAL: NCT03926416
Title: A Randomised, Double-Blind, Double-Dummy, Active and Placebo Controlled Phase I Trial of the Safety, Tolerability and Immunogenicity of the CodaVax Influenza Vaccine
Brief Title: Safety Study of Live Attenuated Influenza Vaccine, CodaVax
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Codagenix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CODA01-001
Record Dates: First submitted 2019-04-18; First posted 2019-04-24 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2019-04

CONDITIONS: Influenza
Keywords: vaccines; live-attenuated vaccine; influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- CodaVax-H1N1, low dose (Experimental): Participants will receive a single dose of either CodaVax (5 x 10^3 PFU in 200 uL) and an intramuscular injection of placebo
  Interventions: Biological: CodaVax-H1N1
- Fluzone (Active Comparator): Participants will receive an intranasal (IN) dose of placebo and an intramuscular (IM) dose of QuadriFlu- Tetravalent Influenza Vaccine (TIV) (Fluzone®)
  Interventions: Biological: Fluzone quadrivalent
- CodaVax-H1N1, high dose (Experimental): Participants will receive a single intranasal (IN) dose of CodaVax-H1N1 (1 x 10^5 PFU in 500 uL)
  Interventions: Biological: CodaVax-H1N1
- Placebo (Placebo Comparator): Leibovitz's L-15 medium (IN) or saline (IM)
  Interventions: Biological: CodaVax-H1N1; Biological: Fluzone quadrivalent

INTERVENTIONS:
Biological: CodaVax-H1N1 — Live-attenuated vaccine against influenza A H1N1, A/California/07/2009
  Arms: CodaVax-H1N1, high dose; CodaVax-H1N1, low dose; Placebo
Biological: Fluzone quadrivalent — Fluzone® (QuadriFlu - TIV), inactivated, quadrivalent influenza vaccine
  Arms: Fluzone; Placebo

SUMMARY:
This study is being conducted to assess the safety, tolerability, and immunogenicity of the CodaVax-H1N1 influenza vaccine as compared to active and placebo controls when administered to healthy adults.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo and active controlled Phase I study is intended to study the effects of a live-attenuated vaccine against influenza A H1N1. Part 1 of this study will enroll 75 participants at a single site. Participants will be randomized in a 2:2:1 ratio to receive one dose each of either CodaVax-H1N1, FluZone quadrivalent, or placebo. This study is conducted during the influenza "off season" in Australia. Part 2 of the study will enroll an 50 additional participants randomized to receive either CodaVax-H1N1 at a higher dose or placebo (40:10).

ELIGIBILITY:
Inclusion Criteria:

* In good health, in the opinion of the Medical Investigator (with or without the Sponsor), with no significant medical history and no clinically significant abnormal findings at screening. Particular attention will be paid to:

  * A drug history identifying any known drug allergies and the presence of drug abuse;
  * Any chronic use of medication(s); and
  * Thorough review of body systems
* Women of child bearing potential (WOCBP) must use highly effective, double contraception from the Screening Visit and up to the Follow-up visit (Day 30 ± 2 days). Double contraception is defined as a condom AND one other form of the following:

  * Established hormonal contraception (with approved oral, injected or depot regimen) for at least 2 months prior to screening
  * Depot or injectable birth control
  * Intrauterine device or intrauterine system in place for at least 2 months prior to screening
  * Documented evidence of surgical sterilization at least 6 months prior to screening visit. i.e., tubal ligation or hysterectomy for women or vasectomy for men (with appropriate post-vasectomy documentation of the absence of sperm in semen) provided the male partner is a sole partner; Males must not donate sperm for at least 70 days post-dose of the last study treatment. Male partners of female participants and female partners of male participants must also use contraception, if they are of childbearing potential.

Women of childbearing potential must have a negative serum pregnancy test at Screening and Day 30. Women not of childbearing potential must be postmenopausal (defined as cessation of regular menstrual periods for at least 12 months), confirmed by FSH level meets the requirement of post-menopausal women if in doubt. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not considered highly effective methods of birth control. Participant abstinence for the duration of the study and 1 month after the last study treatment is acceptable.

* Must be willing to comply with the following conditions to prevent the spread of GMOs according the OGTR Licence (DIR 144):

  1. Hygiene measures intended to prevent interpersonal transmission of study drug must be implemented, including but not limited to frequent handwashing with soap or hand disinfectant, respiratory hygiene and cough etiquette within 7 days following vaccination
  2. Blood, tissue or organs must not be donated within 7 days of vaccination
  3. Severely immunosuppressed persons who require a protective environment are not to be cared for by the participant within 7 days of vaccination
  4. Contact is not to be made with severely immunosuppressed persons who require a protective environment within 7 days of vaccination
  5. All tissues and materials used to collect respiratory secretions are to be sealed in a primary container and placed within a secondary container so that it is not accessible to children or animals for 7 days until it is returned to the study site for disposal, for 7 days within vaccination
* Adequate venous access in the left or right arms to allow collection of a number of blood samples
* No birthmarks, tattoos, wounds or other skin conditions which could reasonably obscure IM injection site reactions
* Able to communicate effectively with study personnel and considered reliable, willing and cooperative in terms of compliance with the protocol requirements
* Participant does not intend to start or change an existing physical conditioning regimen prior to or during the study period
* Participant has voluntarily given written informed consent to participate in the study (prior study entry)
* Participant is available for the duration of the study

Exclusion Criteria:

* Immunodeficiency (including HIV) or autoimmune disorder, or participant is currently taking drugs or was undergoing a form of treatment within 6 weeks prior to study entry that affects the immune system. (Treatment of asthma with low dose corticosteroids equivalent to prednisone <10 mg/day, is permitted).
* Participant is not to have had Guillain-Barre Syndrome
* Received blood or blood products in the 3 months prior to screening
* Received another vaccine within 30 days before screening
* Received another influenza vaccine within 2 years prior to screening
* Participated in another clinical study (involving an investigational product or device) within 60 days before screening (including studies for FluMist®)
* Suffered previous anaphylactic reaction to foods, vaccines, drugs or hymenoptera stings, or has a history of severe allergic reactions (e.g. clinically severe urticaria, asthma)
* Participants with active asthma currently managed by ad lib with inhalers
* Participants with a known egg allergy
* If female, pregnant, planning to become pregnant, or lactating
* Participant has a history of, or current evidence at the time of screening of abuse of alcohol or any drug substance, licit or illicit, or current alcohol consumption is > 4 standard drinks (or equivalent) per day
* History of any psychiatric illness or psychological disorder which may impair the ability to provide written informed consent or participate in the study
* Current or history of significant neurological, cardiovascular, pulmonary (including asthma), hepatic, rheumatic, autoimmune, haematological, metabolic or renal disorder
* Clinically significant abnormal laboratory value at screening as determined by the Investigator
* Unusual dietary habits and excessive or unusual vitamin intake likely, in the opinion of the Investigator, to affect safety pathology parameters
* Participant is seropositive to Human Immunodeficiency Virus (HIV-1 or HIV-2), Hepatitis C Virus (HCV) or HBV.
* Body temperature (oral) ≥38.0ºC or acute illness within 5 days prior to vaccination
* Any skin marking, tattoo or blemish precluding injection site inspection.
* Any other significant finding that, in the opinion of the Investigator, would increase the risk of the individual having an adverse outcome from participating in this study
* Participant is a member of the team or is related or in a dependent relationship with a member of the study team, as defined as the Sponsor or study site personnel

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Number of subjects with solicited local and/or systemic reactions after each vaccination, for each treatment group | 6 days
  Number of volunteers that experience adverse events
Incidence of Adverse Events (AE) | 30 days
  Number of subjects with AEs
Incidence of Serious Adverse Events (SAE) | Days 1-168
  Number of subjects with SAEs

SECONDARY OUTCOMES:
Haemagglutination Inhibition Test (HAI) titre | 30 days post-vaccination
  The percentage of subjects achieving a (HAI) antibody titre ≥ 1:40 determined 30 days post-vaccination as compared to baseline (Day 0, pre-vaccination)
Rate of Seroconversion | 30 days post-vaccination
  The rate of seroconversion, defined as the percentage of subjects with either a pre-vaccination HAI titre < 1:10 and a post vaccination HAI titre > 1:40 or a pre-vaccination HAI titre > or = to 1:10 and a minimum four-fold rise in post-vaccination HAI antibody titre, determined 30 days postvaccination
Cal/09 HAI antibodies | 30 days post-vaccination
  Geometric mean titres (GMT) of anti-A/California/07/2009 (H1N1) HAI serum antibodies 30 days after each vaccination, by treatment group
Mich/15 HAI antibodies | 30 days post-vaccination
  Geometric mean titres (GMT) of anti-A/Michigan/45/2015 (H1N1) antibodies (HAI)
  * Geometric mean fold increase (GMFI) of anti-A/California/07/2009 (H1N1) HAI serum antibodies determined 30 days after each vaccination relative to baseline
  * Geometric mean fold increase (GMFI) of anti-A/Michigan/45/2015 (H1N1) HAI serum antibodies determined 30 days after each vaccination relative to baseline
Increase in anti-Cal/09 antibodies | 30 days post-vaccination
  Geometric mean fold increase (GMFI) of anti-A/California/07/2009 (H1N1) HAI serum antibodies determined 30 days after each vaccination relative to baseline
Increase in anti-Mich/15 antibodies | 30 days post-vaccination
  Geometric mean fold increase (GMFI) of anti-A/Michigan/45/2015 (H1N1) HAI serum antibodies determined 30 days after each vaccination relative to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Paul Griffin, MD, Principal Investigator — Q-Pharm Pty Limited
Locations (1):
- Q-Pharm, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No